CLINICAL TRIAL: NCT01240759
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Study of S-707106 in Subjects With Type 2 Diabetes Mellitus and Inadequate Glycemic Control With Metformin Therapy
Brief Title: Safety and Efficacy of S-707106 in Subjects With Type 2 Diabetes Mellitus and Inadequate Glycemic Control With Metformin Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shionogi (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1010N0921
Record Dates: First submitted 2010-11-11; First posted 2010-11-15 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus; Metformin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- S-707106 Dose A (Experimental): One S-707106 A tablet + 3 Placebo A tablets
  Interventions: Drug: S-707106 Dose A; Drug: Placebo A tablet; Drug: Metformin
- S-707106 Dose B (Experimental): One S-707106 B tablet + 3 Placebo A tablets
  Interventions: Drug: S-707106 Dose B; Drug: Placebo A tablet; Drug: Metformin
- S-707106 Dose C (Experimental): S-707106 Dose C = Four S-707106 B tablets
  Interventions: Drug: S-707106 Dose C; Drug: Metformin
- Metformin (Active Comparator): The standard of care dose of metformin for the individual patient + 3 Placebo A tablets
  Interventions: Drug: Placebo A tablet; Drug: Metformin

INTERVENTIONS:
Drug: S-707106 Dose A — One S-707106 A tablet
  Arms: S-707106 Dose A
Drug: S-707106 Dose B — One S-707106 B tablet
  Arms: S-707106 Dose B
Drug: S-707106 Dose C — Four S-707106 4 X B tablets
  Arms: S-707106 Dose C
Drug: Placebo A tablet — Up to 4 Placebo A tablets
  Arms: Metformin; S-707106 Dose A; S-707106 Dose B
Drug: Metformin — The standard of care dose of metformin for each patient

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of S-707106 co-administered with metformin in subjects with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
Based on the unmet clinical need for more safe and effective type 2 diabetes mellitus therapies, together with the nonclinical efficacy and safety profile of S-707106, Shionogi USA, Inc. is initiating studies to further assess the efficacy, clinical pharmacology and safety profile of S-707106 in preparation for full clinical development as a novel treatment for type 2 diabetes mellitus. It is anticipated that S-707106 will provide clinicians and patients with a new therapeutic option to treat type 2 diabetes mellitus with potential advantages over existing therapy.

ELIGIBILITY:
Main Inclusion Criteria:

* Subjects with type 2 diabetes mellitus receiving a stable dose of metformin for the past 3 months (with no other medication for glycemic control) and who are clinically stable as determined by medical history
* Body mass index (BMI) ≥25.0 and <45.0 (kg/m2) using http://www.bmicalculator.org/ as the BMI calculator
* No clinically significant abnormal laboratory tests as determined by the investigator except Hemoglobin A1c level ≥7.5% and ≤11.0% and C peptide level >1.0 ng/mL

Main Exclusion Criteria:

* Type 1 diabetes mellitus or gestational diabetes mellitus within last 6 months
* Use of any medication for glycemic control other than metformin during the past 3 months or thiazolidinediones within the past year
* Congestive heart failure as defined by New York Heart Association class III or IV
* Fasting glucose >270 mg/dL
* Creatinine clearance is <60 mL/minute
* History of myocardial infarction within the past 3 months, history of clinically significant cardiac arrhythmia, clinically significant hypotension or hypertension, or clinically significant abnormal electrocardiogram as determined by the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2010-10; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline to Week 12 in Hemoglobin A1c (HbA1c) | Baseline and at 12 weeks
  Hemoglobin A1c

SECONDARY OUTCOMES:
Serial pharmacokinetic (PK) assessments | 5 days
  Serial pharmacokinetic sampling at Visit 6 prior to dosing, at Visit 7 prior to dosing and at 0.5, 1, 2, 3, 4, 6, 8 and 24 hours after dosing, at Visit 8, at Visit 9, and Early Termination Visit
Sparse pharmacokinetic assessments | 5 days
  Sparse pharmacokinetic sampling at Visit 6 and Visit 7 prior to dosing, at Visit 6 or Visit 7 one additional post-dose sample, at Visit 8, at Visit 9, and Early Termination Visit
Percent of subjects with Hemoglobin A1c < 7.0% at Week 12 | 12 weeks
  Hemoglobin A1c
Change from Baseline at Week 12 in: Fasting plasma glucose, 1,5-Anhydroglucitol, Fructosamine, Glycoalbumin, C-peptide, Beta-cell function and insulin resistance indices using Homeostatic Model Assessment, and Postprandial glucose test | Baseline and at 12 weeks
  Fasting plasma glucose, 1,5-Anhydroglucitol, Fructosamine, Glycoalbumin, C-peptide, Beta-cell function and insulin resistance indices using Homeostatic Model Assessment, and Postprandial glucose test
Safety assessments | 5-6 months
  Safety will be assessed by monitoring of treatment-emergent adverse events, serious adverse events, treatment-emergent adverse events leading to study drug discontinuation, clinical laboratory evaluations, vital signs, 12-lead electrocardiograms (ECGs), adrenal axis hormones, and treatment-emergent adverse events of hypoglycemia, hyperglycemia, confirmed hypoglycemia or hyperglycemia

CONTACTS AND LOCATIONS:
Overall Officials: Shionogi Clinical Trials Administrator Clinical Support Help Line, Study Director — Shionogi
Locations (1):
- Juno Research, LLC, Houston, Texas, United States